CLINICAL TRIAL: NCT02256995
Title: A Prospective Observational Pilot Study to Test the Feasibility of Smartphone Enabled uChek Urinalysis Device in Bangladesh
Brief Title: uChek Pilot Study for Urinalysis in the Antenatal Care Setting
Acronym: uChekBangla
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maternova Research (Other)
Collaborators: Merck for Mothers (Other); HOPE Foundation for Women and Children of Bangladesh (Unknown)
Responsible Party: Sponsor
Other Study IDs: MATBANG2014
Record Dates: First submitted 2014-09-18; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Preeclampsia; Eclampsia; Pregnancy; Proteinuria
Keywords: Pregnancy; Preeclampsia; Eclampsia; Proteinuria
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pregnant Women (>22 weeks gestation): Biomarkers tracked over 3 antenatal care visits via standard of care (dipstick, manually/visually assessed) and via uChek (automated assessment via computer application)
  Interventions: Device: uChek

INTERVENTIONS:
Device: uChek — The uChek TM urine analyzer is a semi-automated urinalysis system, installed as an application on a smartphone. It makes use of a smartphone's camera to automatically read urine dipsticks.

SUMMARY:
A prospective observational study to test the feasibility of smartphone enabled uChek urinalysis device to detect biomarkers (protein, microalbumin and protein:creatine ratio) in urine, indicative of preeclampsia/eclampsia at over 22 weeks of gestation and assess attitudes of clinicians towards uChek as a new technology for urinalysis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with a gestational age of over 22 weeks and ability to follow pregnancy till delivery.

Exclusion Criteria:

* Study participant is unwilling to take part in study or participants with pathological conditions that restrict them from providing a urine sample without catheterization.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: There are two unique subject populations in this study. One group consists of pregnant women whose urine will be analyzed- hereafter referred to as the Patient Participants. The second group is a cohort of medical professionals who will answer a questionnaire about the usability of the device, relating to the second objective, hereafter referred to as the Medical Staff Participants. The following parameters have been answered in reference to the Patient Participants.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-03 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using uChek for standard urinalysis in an antenatal care (ANC) setting | 6 months
  1. Test the feasibility of using the uChek urinalysis device to detect biomarkers of preeclampsia/eclampsia at over 22 weeks of gestation as compared to using the sites' current urinalysis method. A correlation analysis of the rate of detection of protein in urine between the uChek and the standard visual dipstick test using the quantitative results from the visual dipstick test and uChek results collected at each of three ANC visits.

SECONDARY OUTCOMES:
Impressions and attitudes of healthcare workers re: uChek for urinalysis in ANC | 6 months
  Assess impressions, preferences and attitudes of the clinicians towards the uChek as a tool for urinalysis in antenatal care. A quantitative analysis of questionnaire responses about the usability of the device, including but not limited to:
  * % agree or strongly agree that the uChek is an accurate urinalysis device
  * % reporting that they agree or strongly agree that uChek is easier to use than current method of urinalysis
  * % reporting that they agree or strongly agree that uChek is a suitable technology for a low resource setting

OTHER OUTCOMES:
Feasibility of using uChek for expanded urinalysis panel in ANC | 6 months
  To assess the feasibility of tracking additional biomarkers of conditions affecting pregnant women using urinalysis via the uChek device(glucose for gestational diabetes, nitrites for urinary tract infection, presence of blood, microalbumin for risk of preterm birth, etc.). A quantitative analysis of results of tests for additional biomarkers, detected with the uChek, of conditions affecting pregnant women.

CONTACTS AND LOCATIONS:
Overall Officials: Janardana Sharma, MD, Study Director — Hope Bangladesh
Locations (1):
- Hope Hospital for Women and Children, Cox’s Bāzār, Bangladesh